CLINICAL TRIAL: NCT01649258
Title: A Pilot Study to Evaluate the Efficacy of Fosaprepitant and Granisetron Transdermal System for the Prevention of Acute and Delayed Nausea and Vomiting in Breast Cancer Patients and to Identify Predictors of Response
Brief Title: Fosaprepitant Dimeglumine and Granisetron Transdermal System in Preventing Nausea and Vomiting in Patients With Breast Cancer Undergoing Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-11-5; NCI-2012-01170 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Nausea; Vomiting
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting | interventions — Granisetron; fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive care (antiemetics) (Experimental): Patients receive granisetron transdermal system patch 24-48 hrs before the initiation of chemotherapy. Patients wear the granisetron transdermal system patch for 7 days. Patients receive fosaprepitant dimeglumine IV over 15 minutes on day 1 of chemotherapy. Treatment repeats every 2 or 3 weeks for up to 4 courses in the absence of unacceptable toxicity.
  Interventions: Drug: granisetron transdermal system; Drug: fosaprepitant dimeglumine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: granisetron transdermal system — Given granisetron transdermal system patch
  Other Names: granisetron transdermal patch; Sancuso
Drug: fosaprepitant dimeglumine — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies how well fosaprepitant dimeglumine and granisetron transdermal system work in preventing nausea and vomiting in patients with breast cancer undergoing chemotherapy. Antiemetic drugs may help lessen or prevent nausea and vomiting in patients treated with chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the combination of fosaprepitant (fosaprepitant dimeglumine) and granisetron transdermal system in the prevention of acute and delayed chemotherapy induced nausea and vomiting in breast cancer patients undergoing adjuvant or neoadjuvant chemotherapy.

SECONDARY OBJECTIVE:

I. To evaluate the safety of the combination of fosaprepitant and granisetron transdermal system in breast cancer patients undergoing adjuvan or neoadjuvant chemotherapy.

EXPLORATORY OBJECTIVE:

I. To explore the use of single nucleotide polymorphisms (SNPs) in the 5âhydroxytryptamine-3 (5HT3) and neurokinin-1 (NK-1) receptors as potential markers of efficacy.

OUTLINE: Patients receive granisetron transdermal system patch 24-48 hrs before the initiation of chemotherapy. Patients wear the granisetron transdermal system patch for 7 days. Patients receive fosaprepitant dimeglumine intravenously (IV) over 15 minutes on day 1 of chemotherapy. Treatment repeats every 2 or 3 weeks for up to 4 courses in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed breast cancer scheduled to receive chemotherapy with doxorubicin and cyclophosphamide (adjuvant or neoadjuvant)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Projected life expectancy of at least 3 months
* Provision of informed consent prior to any study-related procedures
* Negative pregnancy test for women of childbearing potential
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000 cells/mm^3
* Hemoglobin >= 9.0g/dL
* Serum creatinine =< 1.5 mg/dl
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 X upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 X upper limit of normal; in patients with bone metastasis and no evidence of liver metastasis and bilirubin =< upper limit of normal an alkaline phosphatase =< 5 ULN will be allowed
* Serum bilirubin =< 1.0 mg/dL
* No other concomitant therapy directed at the cancer is allowed

Exclusion Criteria:

* Allergy or intolerance to 5HT3 or NK-1 antagonists and dexamethasone
* Use of another antiemetic agent (5HT3 antagonists, phenothiazines, butyrophenones, cannabinoids, metoclopramide, or corticosteroids) within 72 hours prior to day 1 of the study
* Use of anticoagulant agent (Warfarin, Coumadin, Jantoven, Marevan, Lawarin, Waran, or Warfant)
* An episode of vomiting or retching within 24 hours before the start of the initial treatment with chemotherapy
* Severe concurrent illness other than neoplasia
* Gastrointestinal obstruction or an active peptic ulcer
* Patients who are pregnant or breast feeding because aprepitant may be harmful to the developing fetus and newborn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete response, defined as no emesis and no use of rescue medication in acute phase (within first 24 hours of treatment) | Within the first 24 hours of treatment
  The complete response rate with the exact 95% confidence intervals (CIs) will be calculated. The associations between the complete response rate and patient characteristics and biomarkers will be examined using Fisherâs exact test or Mann-Whitney U test whenever appropriate.
Proportion of patients with complete response, defined as no emesis and no use of rescue medication in delayed phase (within 2-4 days of treatment) | Up to day 4
  The complete response rate with the exact 95% CIs will be calculated. The associations between the complete response rate and patient characteristics and biomarkers will be examined using Fisherâs exact test or Mann-Whitney U test whenever appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States